CLINICAL TRIAL: NCT00272662
Title: A Phase 2, Open-Label, Multi-Center Dose Escalation Study of the Safety, Pharmacodynamics, and Pharmacokinetics of Subcutaneously Administered Peginesatide in Anemic Cancer Patients Receiving Chemotherapy
Brief Title: Study of Subcutaneously Administered Peginesatide in Anemic Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-05; 2005-003354-10 (EudraCT Number)
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Chemotherapy Induced Anemia; Cancer
Keywords: anemia; cancer; chemotherapy; chemotherapy induced anemia; CIA; hemoglobin; Hb; Hgb; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Neoplasms; Anemia | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Peginesatide starting dose of 0.1 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 3 weeks (Q3W) for a total of 4 doses.
  Interventions: Drug: peginesatide
- Cohort 2 (Experimental): Peginesatide starting dose of 0.15 mg/kg administered SC Q3W for a total of 4 doses.
  Interventions: Drug: peginesatide
- Cohort 3 (Experimental): Peginesatide starting dose of 0.2 mg/kg administered SC Q3W for a total of 4 doses.
  Interventions: Drug: peginesatide
- Cohort 4 (Experimental): Peginesatide starting dose of 0.05 mg/kg administered SC Q3W for a total of 4 doses.
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide
  Other Names: Omontys; Hematide; AF37702 Injection

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacodynamics (PD), and pharmacokinetics (PK) of multiple subcutaneously administered injections of peginesatide in anemic cancer participants receiving chemotherapy.

DETAILED DESCRIPTION:
This was a Phase 2, open-label, multi-center, sequential dose finding study with up to 6 treatment cohorts receiving chemotherapy with 15 participants per cohort. The primary objective of this study was to determine the dose of peginesatide administered every 3 weeks (Q3W) by subcutaneous injection associated with a hemoglobin increase of ≥ 1 g/dL in ≥ 50% of anemic cancer participants receiving chemotherapy at 9 weeks following the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local, and national guidelines
* Males or females ≥ 18 and ≤ 80 years of age; pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice a highly effective method of birth control for at least 2 weeks prior to study start, and must be willing to continue practicing birth control for at least 4 weeks after the last dose of study drug. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence (only acceptable if practiced as a life-style and not acceptable if one who is sexually active practices abstinence only for the duration of study) or vasectomized partner
* Participants with histologically confirmed solid tumor malignancy or lymphoma who are scheduled to receive at least 9 weeks of cyclic myelosuppressive chemotherapy while on study
* Hemoglobin value of ≥ 8 and < 11 g/dL within 1 week prior to administration of study drug.
* ECOG Performance Status of 0-2
* One reticulocyte hemoglobin content (CHr) > 29 picograms within 4 weeks prior to study drug administration.
* One transferrin saturation ≥ 15% within 4 weeks prior to study drug administration.
* One serum or red cell folate level above the lower limit of normal within 4 weeks prior to study drug administration
* One vitamin B12 level above the lower limit of normal within 4 weeks prior to study drug administration
* One absolute neutrophil count ≥ 1.0 x 10^9/L within 1 week prior to administration of study drug
* One platelet count ≥ 75 x 10^9/L within 1 week prior to administration of study drug
* Life expectancy > 6 months.

Exclusion Criteria:

* Treatment with any erythropoiesis stimulating agent (ESA) in the past 90 days
* History of failure to respond to ESA treatment
* Known antibodies to other ESAs or history of pure red cell aplasia (PRCA)
* Acute or chronic leukemia, myelodysplastic syndrome (MDS), or multiple myeloma
* Any previous or planned radiotherapy to more than 50% of either the pelvis or spine
* Known intolerance to parenteral iron supplementation
* Red blood cell transfusion within 4 weeks prior to study drug administration
* Known hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all types, etc.)
* Known hemolysis
* History of pulmonary embolism or deep venous thrombosis (DVT) in the previous 2 years or current therapeutic doses of anticoagulants
* Known blood loss as a cause of anemia
* Uncontrolled, or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times the upper limit of normal; AST or ALT > 5 times the upper limit of normal if liver metastases are present.
* Creatinine > 175 micromoles per liter (µmol/L)
* History of bone marrow or peripheral blood cell transplantation
* Pyrexia/fever of ≥ 39 °C within 48 hours prior to study drug administration
* Poorly controlled hypertension, per the Investigator's judgment, within 4 weeks prior to study drug administration (e.g., systolic ≥ 170 mm Hg or diastolic ≥ 100 mm Hg on repeat readings)
* Epileptic seizure in the 6 months prior to study drug administration
* Advanced chronic congestive heart failure - New York Heart Association Class IV
* High likelihood of early withdrawal or interruption of the study
* Anticipated elective surgery during the study period
* History of multiple drug allergies
* Exposure to any investigational agent within 1 month prior to administration of study drug or planned receipt during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a hemoglobin increase of ≥ 1 gram per deciliter (g/dL) at 9 weeks following Dose 1 | Week 9 post Dose 1

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | 13 Weeks
Time to achieve hemoglobin increase ≥ 1 g/dL from baseline | Baseline to Week 13
Proportion of participants with a hemoglobin response | 13 Weeks
Pharmacokinetic parameters | 13 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Affymax, Study Director — Affymax, Inc
Locations (10):
- Czechia (4):
  - Research Facilities, Brno
  - Research Facility, Hradec Králové
  - Research Facility, Olomouc
  - Research Facility, Příbram
- Poland (5):
  - Research Facility, Gdansk
  - Research Facilities, Krakow
  - Research Facility, Lodz
  - Research Facility, Poznan
  - Research Facility, Szczecin
- Research Facilities, London, United Kingdom